CLINICAL TRIAL: NCT04473404
Title: Evaluation of the Effect of an Oral Probiotic on Oral Bacteria and Malodor
Brief Title: Effect of a Probiotic Water on Oral Health in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dose Biosystems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DB001-2020
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-07

CONDITIONS: Oral Bacteria; Halitosis
Keywords: Probiotic; Oral microbiome
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic - low dose (Experimental): Powdered probiotic with a carrier.
  Interventions: Dietary Supplement: Streptococcus salivarius DB-B5 - 2 billion CFU/day
- Probiotic - high dose (Experimental): Powdered probiotic with a carrier.
  Interventions: Dietary Supplement: Streptococcus salivarius DB-B5 - 10 billion CFU/day
- Placebo (Placebo Comparator): Carrier only.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius DB-B5 - 2 billion CFU/day — The participants (n=15) will consume sachets containing Streptococcus salivarius DB-B5 (at 1 billion CFU/sachet) dissolved in water twice daily for 4 weeks.
  Arms: Probiotic - low dose
Dietary Supplement: Streptococcus salivarius DB-B5 - 10 billion CFU/day — The participants (n=15) will consume sachets containing Streptococcus salivarius DB-B5 (at 5 billion CFU/sachet) dissolved in water twice daily for 4 weeks.
  Arms: Probiotic - high dose
Other: Placebo — The participants (n=15) will consume sachets containing a placebo (probiotic carrier) twice daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of consuming a probiotic on salivary, plaque, and tongue bacteria, as well as oral malodor (bad breath). Healthy volunteers will consume a probiotic powder, or a placebo powder, that is dissolved in water for 4 weeks.

DETAILED DESCRIPTION:
The oral cavity houses one of the most diverse microbiota in the human body. There are nearly 800 unique oral bacterial species identified with more species expected to be added with further sampling and identification. As with microbiota of other sites in the body, a balanced oral microbiota is essential to maintaining the health of the human host. Streptococcus salivarius is a pioneer species that colonizes the human oral cavity from birth, and remains a predominant member of the commensal microbiota throughout life. The commensal microbiota provides protection against pathogenic species associated with conditions such as dental caries, periodontal disease, and oral malodor (halitosis). This randomized, double-blind, placebo-controlled study is conducted to investigate the effect of a Streptococcus salivarius DB-B5 strain on oral bacteria levels and halitosis. Doses of 2 billion and 10 billion colony forming units (CFU) per day are tested.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 to 65 years of age and in good general health and good oral health (no active or uncontrolled diseases or conditions).
2. Presence of at least 20 natural teeth, excluding third molars.
3. Read and sign the Research Subject Information and Consent Form.
4. Have an OralChroma reading ≥ 125 ppb hydrogen sulfide (H2S) gas, volatile sulfur compound (VSC) (at least 8-12 hours after eating or drinking or oral hygiene) at Baseline.
5. Willingness to use the assigned products according to instructions, attend scheduled appointments, and likelihood of completing the study.
6. Males and females with reproductive potential agree to use medically acceptable contraception, as determined by the investigator, for the duration of the study and 30 days after study completion and attest to having used it for three months prior to screening.
7. Females of child-bearing potential agree to submit to a urine pregnancy test at screening and at the end of the study.

Exclusion Criteria:

1. Fewer than 20 natural, uncrowned teeth.
2. Active or chronic dental disease.
3. Self-reported dry mouth (xerostomia) by questionnaire.
4. Have had or used any of the following in the past three months: antibiotic treatment, a dental cleaning, mouthrinse.
5. Regular use of probiotic supplements or regular consumption of probiotic rich foods such as yoghurt or kefir in the past month.
6. Require antibiotic prophylaxis for dental or any treatment.
7. Removable or fixed dental appliances (no implants; crowns allowed if subject has at least 20 uncrowned teeth)
8. Pregnant or planning to become pregnant during the study period, or breastfeeding.
9. Uses tobacco products (including smokeless, vaping, and nicotine chewing gums/sprays/lozenges).
10. Chronic or acute illness such as heart disease, diabetes, cancer, autoimmune condition or HIV that could impact outcome of the study in the opinion of the investigator.
11. Use of a dental product or is on a medication/treatment that could impact outcome of the study in the opinion of the investigator.
12. Is unwilling or unable to provide informed consent and follow study procedures.
13. Has participated in any clinical study within 30 days.
14. Clinical site personnel or relative or partner of clinical site personnel.
15. Any other condition or situation that may increase the risk associated with study participation or may interfere with the study results in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Oral bacteria levels in saliva and plaque | 4 weeks
  Change in the levels of the following bacteria in the saliva, and in samples of supra- and subgingival plaque: Streptococcus salivarius (total), Streptococcus salivarius DB-B5 (probiotic strain), Streptococcus mutans and Porphyromonas gingivalis.
Oral bacteria levels on the tongue | 4 weeks
  Change in the levels of the following bacteria in back-of-tongue samples: Tannerella forsythia, Prevotella (total), Streptococcus salivarius (total) and Streptococcus salivarius DB-B5 (probiotic strain).
Oral malodor | 4 weeks
  Change in OralChroma malodor readings.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L. Milleman, DDS, MPA, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States